CLINICAL TRIAL: NCT00574951
Title: A Phase II Evaluation of AMG 706 (IND # 79,697) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: AMG 706 in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped for severe toxicity causing concern for patients
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170L; GOG-0170L; AMGEN-20060747
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Results first posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2015-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: fallopian tube cancer; recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — motesanib diphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMG 706 (Experimental): AMG 706 daily
  Interventions: Drug: motesanib diphosphate

INTERVENTIONS:
Drug: motesanib diphosphate

SUMMARY:
RATIONALE: AMG 706 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well AMG 706 works in treating patients with persistent or recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the activity of AMG 706, in terms of the frequency of patients with progression-free survival for at least 6 months after initiating therapy or with an objective tumor response, in patients with persistent or recurrent ovarian epithelial, fallopian tube, or primary peritoneal carcinoma.

Secondary

* To determine the frequency and severity of adverse events as assessed by CTCAE v3.0.
* To characterize the distribution of the progression-free and overall survival of these patients.

OUTLINE: This is a multicenter study.

Patients receive oral AMG 706 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal carcinoma

  * Recurrent or persistent disease
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan

  * Must have at least one "target lesion" that can be used to assess response, as defined by RECIST criteria

    * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented OR a biopsy is obtained to confirm persistent disease ≥ 90 days following completion of radiotherapy
* Must have received one prior platinum-based chemotherapeutic regimen containing carboplatin, cisplatin, or another organoplatinum compound for management of primary disease

  * Initial treatment may have included high-dose therapy, consolidation therapy, or extended therapy administered after surgical or non-surgical assessment
  * One additional cytotoxic regimen for management of recurrent or persistent disease allowed
  * Patients must have a platinum-free interval of < 12 months, have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Ineligible for a higher priority GOG protocol
* No pleural effusion or ascites causing grade 2 or greater dyspnea
* No history of uncontrolled CNS metastases

  * Patients with a history of CNS metastases must have their disease controlled by radiotherapy and/or surgery; have at least two imaging scans following treatment (that were no less than 30 days apart) showing no progression of any lesions and no new lesions; and be clinically stable off corticosteroids for ≥ 14 days prior to study randomization

PATIENT CHARACTERISTICS:

* GOG performance status (PS) 0-2* NOTE: *Patients who have received 2 prior regimen must have a GOG PS of 0-2 and patients who have received 2 prior regimens must have a GOG PS of 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Urine protein < 30 mg/dL by urinalyses or ≤ 1+ by urine dipstick (unless quantitative protein is < 500 mg by 24-hour urine collection)
* Bilirubin ≤ 1.5 times ULN (< 3 times ULN in patients with UGT1A1 promoter polymorphism [i.e., Gilbert syndrome] confirmed by genotyping or Invader® UGT1A1 Molecular Assay)
* AST and ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 2 times ULN (5 times ULN if liver or bone metastases are present)
* PTT normal
* INR ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow oral medications
* Cardiac ejection fraction normal
* No sensory and motor neuropathy > grade 2
* No other invasive malignancies within the past 5 years, except nonmelanoma skin cancer or other specific malignancies
* No bleeding diathesis or hypercoagulopathy within the past 14 days
* No arterial or venous thrombosis within the past 12 months
* None of the following within the past 12 months:

  * Myocardial infarction
  * Cerebrovascular accident
  * Transient ischemic attack
  * Grade 2 or greater peripheral vascular disease
  * Percutaneous transluminal coronary angioplasty/stent
  * Congestive heart failure
  * Ongoing arrhythmias requiring medication
  * Unstable angina
* No average systolic blood pressure ≥ 150 mm Hg and average diastolic blood pressure ≥ 90 mm Hg

  * Patients with hypertension that is stable on a current dose of anti-hypertensives are eligible
* No history of impaired cardiac status (e.g., severe heart disease, cardiomyopathy, or congestive heart failure)
* No psychiatric, addictive, or other kind of disorder that would compromise the ability of the patient to give written informed consent
* No open wounds, ulcers, or fractures
* No active infection requiring antibiotics (with the exception of uncomplicated UTI)
* No known HIV, hepatitis B, or hepatitis C positivity
* No known hypersensitivity to AMG 706

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered form prior surgery, radiotherapy, or chemotherapy
* At least 1 week since prior hormonal therapy for the malignant tumor

  * Concurrent hormone replacement therapy allowed
* At least 3 weeks since other prior therapy directed at the malignant tumor, including biologic or immunologic agents (i.e., small molecules or murine monoclonal antibodies)
* At least 12 weeks since prior chimeric, human, or humanized monoclonal antibodies
* More than 30 days since prior investigational therapy
* More than 12 weeks since prior bevacizumab
* More than 30 days since prior VEGFR-targeted therapy, including, but not limited to, any of the following:

  * SU5416
  * SU6668
  * Sunitinib malate
  * Vandetanib
  * Vatalanib
  * AZD2171
  * AEE 788
  * Sorafenib
* More than 28 days since prior major surgery
* More than 14 days since prior minor surgery, including open breast biopsy
* More than 7 days since prior core needle biopsy or placement of a central venous access device (including portion, tunneled, or non-tunneled catheters)
* No prior cancer treatment that would contraindicate study therapy
* No prior therapy AMG 706
* No prior chemotherapy for any abdominal or pelvic tumor other than for the treatment of ovarian, fallopian tube, or primary peritoneal cancer

  * Prior adjuvant chemotherapy for localized breast cancer allowed provided it was completed > 3 years ago, and the patient remains free of recurrent or metastatic disease
* No prior non-cytotoxic chemotherapy for management of recurrent or persistent disease
* No prior radiotherapy to any portion of the abdominal cavity or pelvis other than for the treatment of ovarian, fallopian tube, or primary peritoneal cancer

  * Prior radiotherapy for localized cancer of the breast, head and neck, or skin allowed provided it was completed > 3 years ago, and the patient remains free of recurrent or metastatic disease
* No concurrent coumadin-type anticoagulants, including warfarin, at doses > 1 mg/day

  * Concurrent low molecular weight heparin or low dose warfarin (i.e., ≤ 1 mg daily) for prophylaxis against central venous catheter thrombosis is allowed
* No other concurrent investigational or antineoplastic agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell J. Schilder, MD, Study Chair — Fox Chase Cancer Center
Locations (19):
- United States (19):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - University of Illinois Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Harrington Cancer Center, Amarillo, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 12/10/2007 and closed to accrual on 4/22/2008.
Groups:
- AMG 706: AMG 706 125 mg PO daily continuously (one cycle is 28 days) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | AMG 706
Started | 23
Completed (Eligible and treated patients.) | 22
Not Completed | 1
Not completed — Ineligible - improper prior treatment | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | AMG 706
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.6)
Age, Customized [Count of Participants; unit: Participants]
  Age at study entry: 50-59 years | 7
  Age at study entry: 60-69 years | 9
  Age at study entry: 70-79 years | 5
  Age at study entry: 80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI every other cycle for the first 6 months; then every 3 months thereafter; and at any other time if clinically indicated up to 5 years.
Population: Eligible and treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 706
Number analyzed (Participants) | 22
Participants
  Partial response | 1
  Complete response | 0

2. Primary Outcome: Progression-free Survival (PFS) at 6 Months
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions. In this study, time of progression could not be validly collected due to the study being prematurely closed secondary to severe neurological adverse events seen in 4 patients,
Time Frame: CT scan or MRI every other cycle for the first 6 months
Population: Time of progression could not be validly collected due to the study being prematurely closed due to severe neurological adverse events, thus 6-month PFS cannot be presented. For safety reasons, most patients (16/22) were taken off study drug prior to progression (or AE), and follow-up for progression after coming off study was not collected.
Arm/Group | AMG 706
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Overall Survival (OS)
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 706
Number analyzed (Participants) | 22
months | 13.1 [8.1 to NA] — Not available because data was not sufficiently mature at the time of analysis to calculate the estimate. Won't become available because study was terminated for toxicity

4. Secondary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: Number of participants with a maximum grade of 3 or higher during the treatment period.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 706
Number analyzed (Participants) | 22
Participants
  Cardiac | 2
  Gastrointestinal | 5
  Hepatobiliary | 1
  Metabolic | 4
  Muskuloskeletal | 1
  Other Neurological | 4
  Pain | 1
  Pulmonary | 1
  Death, Not CTC coded | 1

5. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions. In this study time of progression could not be validly collected due to the study being prematurely closed, secondary to severe neurological adverse events seen in 4 patients, and thus progression-free survival (PFS) cannot be presented. For safety reasons, most patients (16/22) were taken off study drug prior to progression (or AE),
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; then every 3 months thereafter; and at any other time if clinically indicated, up to 5 years
Population: Study Analysis aborted due to severe toxicities. Estimates not calculated. Follow up for progression after coming off study was not collected in a manner that yields time to time to progression data.
Arm/Group | AMG 706
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | AMG 706
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 706 (N=22)
Hypertension (Cardiac disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 706 (N=22)
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 7
Hemoglobin (Blood and lymphatic system disorders) | 11
Palpitations (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 9
Weight Loss (General disorders) | 2
Fatigue (General disorders) | 15
Rash (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 3
Heartburn (Gastrointestinal disorders) | 2
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Anorexia (Gastrointestinal disorders) | 6
Dehydration (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 9
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 2
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 1
Ast (Metabolism and nutrition disorders) | 7
Creatinine (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alt (Metabolism and nutrition disorders) | 5
Alkaline Phosphatase (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Nervous system disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Cns Ischemia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 6
Neuropathy-Motor (Nervous system disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Head/Headache (General disorders) | 13
Pain: Extremity-Limb (General disorders) | 4
Pain: Back (General disorders) | 4
Pain: Joint (General disorders) | 2
Pain: Bone (General disorders) | 1
Pain: Stomach (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 4
Pain: Skin (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less